CLINICAL TRIAL: NCT06600152
Title: A Randomized, Open-label, Investigational Safety Evaluation of the Microporous Annealed Particle (MAP) Wound Matrix (TT101) Device as a Volumetric Biomaterial Scaffold Applied to Clean Wounds After Skin Cancer Surgery With Mohs Micrographic Surgery (MMS) Compared to Control.
Brief Title: Safety of Microporous Annealed Particle (MAP) Wound Matrix in Patients With Clean Surgical Wounds.
Acronym: MOSAIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tempo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT-CLN-004-03
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Wound Heal
MeSH Terms: interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Intervention Model Description: 2:1 randomization model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Microporous Annealed Particle (MAP) Wound Matrix (Experimental): The Microporous Annealed Particle (MAP) Wound Matrix device will be topically applied to the wound immediately following Mohs micrographic surgery (MMS).
  Interventions: Device: MAP Wound Matrix
- Hydrocolloid dressing (DuoDerm) (Active Comparator): A hydrocolloid (DuoDerm) will be topically applied to the wound immediately following Mohs micrographic surgery.
  Interventions: Device: DuoDerm

INTERVENTIONS:
Device: MAP Wound Matrix — The MAP Wound Matrix is indicated for the management of full thickness wounds, including surgical sites, donor skin graft sites, wound dehiscence, lacerations, and draining wounds. The application of MAP Wound Matrix will occur immediately after Mohs surgery once hemostasis has been achieved
  Arms: Microporous Annealed Particle (MAP) Wound Matrix
Device: DuoDerm — DuoDerm is a hydrocolloid dressing will be topically applied to the wound immediately following Mohs surgery according to the manufacturer's instructions.
  Arms: Hydrocolloid dressing (DuoDerm)

SUMMARY:
A randomized, open-label, investigational safety evaluation of the Microporous Annealed Particle (MAP) Wound Matrix (TT101) device as a volumetric biomaterial scaffold applied to clean wounds after skin cancer surgery with Mohs micrographic surgery (MMS) compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo the written informed consent process prior to enrollment in this study.
* At least 22 years of age at screening.
* Has non-melanoma skin cancer and be scheduled for skin cancer surgery with Mohs micrographic surgery on a location suitable for secondary intention healing.
* Resulting surgical wound after Mohs micrographic surgery must be at least 1 cm and no more than 4 cm in diameter (or surface area of at least 0.8 cm2 and no more than 12.6 cm2).
* Resulting surgical wound after Mohs micrographic surgery must be full thickness.
* Willing to return for all required follow-up visits.
* Willing to follow the instructions of the Principal Investigator.

Exclusion Criteria:

_ Has a confirmed diagnosis of clinically significant peripheral neuropathy.

* Has uncontrolled Type I or Type II diabetes and HbA1c values greater than 8.0% within the last 6 months.
* Has a known infection in the area of the Mohs micrographic surgery.
* Has a known allergy to any of the components of the TT101 Device.
* Is an active daily cigarette smoker.
* Is pregnant or lactating.
* Is a woman of child-bearing potential who is unwilling to avoid pregnancy or use an appropriate form of birth control (adequate birth control methods are defined as: topical, oral, implantable, or injectable contraceptives; spermicide in conjunction with a barrier such as a condom or diaphragm; IUD; or surgical sterilization of partner).
* Has clinical evidence of Peripheral Vascular Disease (PVD) in the form of grade 2 pitting Edema or higher.
* Has been diagnosed with a surgical or wound site infection within the last 6-months.
* Has been diagnosed with chronic ulcer or wound within the last 12- months.
* Has a remote active infection concurrent with having the Mohs micrographic surgery.
* Per Investigator's discretion the subject is not appropriate for inclusion in the trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse device effects in the treatment group compared to the control group. | Week 0 (treatment) up to Week 24 (End of Study)
  Incidence of serious adverse device effects (SADE) (including delays in wound healing and surgical site infections) in subjects treated with MAP Wound Matrix, compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Quach, BS, Study Director — Tempo Therapeutics
Locations (3):
- United States (3):
  - Cal Coast Dermatology, Encino, California
  - Laser and Skin Surgery Center of Indiana, Indianapolis, Indiana
  - Studies in Dermatology, Cypress, Texas

IPD SHARING:
Plan to Share IPD: Yes